CLINICAL TRIAL: NCT03389360
Title: Evaluation of Procalcitonin (PCT) as a Marker of Infection Post Living Donated Liver Transplant
Status: Completed | Type: Observational
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, Fellow of intensive care medicine, National Hepatology & Tropical Medicine Research Institute
Other Study IDs: NHTMRI
Record Dates: First submitted 2017-12-25; First posted 2018-01-03 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Liver Transplant Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: procalcitonin — assessing the frequency of rising procalcitonin associated with infectious complications in immunosuppressed LDLTRx.

SUMMARY:
, the study aimed at assessing the frequency of rising procalcitonin associated with infectious complications in immunosuppressed LDLTRx.

DETAILED DESCRIPTION:
All patients transferred from operative theatre to ICU will be sedated, intubated & ventilated. They will receive empiric antimicrobial prophylaxis upon admission & early immunosuppression according to the clinical practice guidelines in our center, (Appendix 1).

Preoperative patients' demographic data will be obtained. Model for end-stage liver disease (MELD) prior transplant, the primary cause of liver transplant.

Operative & anesthetic details; operation time, units of blood, blood products transfusion, ischemic time, type of preservatives used, back table procedures, extra-hepatic procedure & graft to recipient weight ratio will be recorded.

Postoperative patient evaluation will include; Sequential Organ Failure Assessment (SOFA) on admission & /48h. Hemodynamic monitoring will include hourly measurement of heart rate, mean arterial pressure (MAP), temperature, central venous pressure (CVP), arterial oxygen saturation (SaO2), daily total volume of fluid infused, urine output, fluid balance daily, blood gases / 6h & daily mean values will be recorded till hospital discharge.

Routine laboratory workup includes biochemical markers of liver, kidney function and hematological parameters (complete blood count & coagulation profile).

Patient evaluation for infection will be done through scheduled measurements of PCT every other day during ICU stay & upon needed during the hospital stay. Other markers of infections will be measured till hospital discharge as C-reactive protein (CRP) every other day, daily total leukocyte count (TLC) & band cells %.

Microbiological evidence of infection will be confirmed by cultures that will be regularly sampled every other day during ICU stay & upon any clinical or laboratory biomarker suggestive of infection.

Management of suspected infection; when PCT value rising with clinical, radiological &/or laboratory evidence of infection (TLC, CRP, band%), culture from suspected site of infection will be withdrawn. If the source of infection is not evident, cultures from; blood, urine, sputum, surgical wound, drain & nasal swab will be withdrawn & empiric antimicrobial against gram +ve bacteria will be initiated. While the management of proven infection will be culture based antimicrobial initiation.

ELIGIBILITY:
Inclusion Criteria:

* including adult patients aged ≥18 years old who are recipients for living donated liver transplantation (LTx) at the Department of Liver Transplant of National Hepatology & Tropical Medicine Research Institute (NHTMRI), between January 2014 and January 2018 & with no contraindications for early immunosuppression.

Exclusion Criteria:

* Patients will be excluded from the study if they are readmitted or had primary graft nonfunction.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients aged ≥18 years old who are recipients for living donated liver transplantation (LTx)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
frequency of rising procalcitonin associated with infectious complications in immunosuppressed LDLTRx. | average two weeks during hospital stay
  value of procalcitonin to diagnose infection in early post liver transplant period

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided